CLINICAL TRIAL: NCT05307354
Title: The Effectiveness of Tibial Nerve Mobilization in Patients With Tarsal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: KutahyaHSUtibialnerve
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-03

CONDITIONS: Nerve Compression Syndromes; Neuropathic Pain
MeSH Terms: conditions — Nerve Compression Syndromes; Neuralgia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerve Mobilization Group (Experimental): Tibial nerve mobilization in addition to foot-ankle joint range of motion exercises
  Interventions: Other: Tibial Nerve Mobilization; Other: Foot-ankle range of motion exercises
- Control group (Active Comparator): Only joint range of motion exercises
  Interventions: Other: Foot-ankle range of motion exercises

INTERVENTIONS:
Other: Tibial Nerve Mobilization — The person performing tibial nerve mobilization will start mobilization by keeping the lower extremity in a horizontal position, with the patient's hip and knee in 45° flexion and ankle in neutral position. Then, in order to mobilize the tibial nerve better, the patient will bring the patient's toes to the extension position, the ankle to the dorsiflexion and eversion position, and the knee joint to the extension to provide appropriate stabilization. Finally, while the patient is in this position, mobilization will be completed by plantar flexion of the distal ankle and flexion of the toes to allow the nerve to slide further distally. This mobilization technique will be performed by an experienced physician/physiotherapist twice a week for 4 weeks, and the patients will be given 5 sets of 10 cycles with a 1-minute rest period in each set.
  Arms: Nerve Mobilization Group
Other: Foot-ankle range of motion exercises — In exercise program, foot-ankle joint range of motion exercises will be given. In our study, all exercises will be explained and performed once under the supervision of a physiotherapist, and then the participants will be asked to do all exercises with 10 repetitions, 3 times a day, for four weeks, without the supervision of a physiotherapist.

SUMMARY:
This randomized, clinical, single-blinded, controlledstudywasinitiallyplannedtoinclude 35 patients diagnosed with tarsal tunnel who applied to Kütahya Health Sciences University, Evliya Çelebi Training and Research Hospital, Physical Medicine and Rehabilitation outpatient clinic.Patients aged 20-55 years who were diagnosed with tarsal tunnel syndrome by electromyography (EMG) in the last 6 months were included in the study. The patients were randomized into two groups using the computer-assisted randomization method. Tibial nerve mobilization and foot-ankle range of motion exercises will be given to the study group, and only foot-ankle joint range of motion exercises will be given to the control group. All the patients were evaluated with the Visual Analog Scale (VAS), Foot Functional Index (FFI), Neuropathic Pain QuestionnaireN (NPQ) and Tibial Nerve ultrasonography before the intervention and at the fourth week of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-55 years who were diagnosed with tarsal tunnel syndrome by electromyography (EMG) in the last 6 months were included in the study.

Exclusion Criteria:

* Have a systemic inflammatory disease
* Presence of a cognitive disorder, receiving psychotherapy or any psychiatric treatment, disease affecting the central nervous system
* Being illiterate
* Having hearing, vision problems
* History of foot and ankle surgery
* Any pathology that may cause pain in the foot joint diagnosed on physical examination
* Inadequate function of any extremity that would prevent exercise
* The presence of a balance disorder or a disease that can disrupt the balance
* Diagnosis of advanced cardiac or lung disease for which exercise would be contraindicated

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | Change from Baseline at 4th weeks
  VAS, a scale consisting of a single line of 10 cm, was used to evaluate pain severity.
Evaluation of the tibial nerve with ultrasonography | Change from Baseline at 4th weeks
  Bilateral tibial nerve US evaluation using a 6-18 Mhz linear probe (Mindray-UMT 200, USA) will be performed by another clinician experienced in musculoskeletal ultrasonography and blind to the clinical evaluation findings of patients.
Tinel's Sign | Change from Baseline at 4th weeks
  It is performed by lightly tapping (percussing) over the nerve to elicit a sensation of tingling or "pins and needles" in the distribution of the Tibial nerve. The Tinel sign is the tingling or prickling sensation elicited by the percussion of an injured nerve trunk at or distal to the site of the lesion. The test is positive when a tingling or prickling sensation is felt in the distribution of the Tibial nerve.

SECONDARY OUTCOMES:
Foot Function Index | Change from Baseline at 4th weeks
  The severity of foot pain was scored with 23 items measuring the degree of difficulty in performing various functional activities due to foot problems and activity limitations due to foot problems. Turkish validity and reliability of the questionnaire was determined by Yalıman et al.
Neuropathic pain questionnaire | Change from Baseline at 4th weeks
  Neuropathic pain questionnaire consists of 12 questions. Of the 12 questions, 10 are related to the character of the pain while two questions are related to sensitivity changes.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Akdeniz LEBLEBİCİER, MD, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Yes